CLINICAL TRIAL: NCT00389181
Title: A Randomized Trial of Unruptured Brain Arteriovenous Malformations
Brief Title: A Randomized Trial of Unruptured Brain AVMs
Acronym: ARUBA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jay Preston Mohr, Daniel Sciarra Professor of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAB6286; U01NS051566 (NIH); U01NS051483 (NIH)
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Arteriovenous Malformations, Cerebral
Keywords: Unruptured brain arteriovenous malformation; AVM; BAVM; Stroke; Intracranial Hemorrhage
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Stroke; Intracranial Hemorrhages | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical management (Experimental): Patients with unruptured BAVMs will receive symptomatic medical management alone.
  Interventions: Other: Medical management
- Interventional therapy (Active Comparator): Patients with unruptured BAVMs will receive symptomatic medical management with invasive therapies (any combination of surgery, endovascular embolization, or radiotherapy).
  Interventions: Procedure: Interventional therapy; Other: Medical management

INTERVENTIONS:
Procedure: Interventional therapy — All interventional procedures are standard of care for the treatment of AVMs. They are not experimental. A patient randomized to interventional therapy is expected to begin interventional therapy within 3 months following randomization. Interventional therapy consists of endovascular attempts at occlusion of the nidus and feeding vessels, coiling or microsurgery for feeding artery aneurysms, microsurgery for BAVM itself, and radiosurgery, these alone or in various combinations and timings.
  Arms: Interventional therapy
Other: Medical management — Patients participating in the trial will receive the best medical management possible for the disorder being tested in the trial and for any general medical illnesses they are demonstrated to have. One important consideration in the medical management of patients in this trial is stroke risk factor reduction.

SUMMARY:
The purpose of this study is to determine if medical management is better than invasive therapy for improving the long-term outcome of patients with unruptured brain arteriovenous malformations.

DETAILED DESCRIPTION:
Brain arteriovenous malformations (BAVMs) are an infrequent but important cause of stroke, particularly in a young population. Current invasive treatment strategies are varied and include endovascular procedures, neurosurgery, and radiotherapy. All of these treatments are administered on the assumption that they can be achieved at acceptably minor complication rates, decrease the risk of subsequent hemorrhage, and lead to better long-term outcomes.

Recent data from the literature comparing initial presentation and outcome for patients with ruptured and unruptured BAVMs have raised the possibility that such elective invasive treatment for unruptured BAVMs may yield worse outcomes than managing patients symptomatically with therapy. Unfortunately, no controlled clinical trials have yet been undertaken for management of unruptured BAVMs to address these concerns. Therefore, the goal of this randomized controlled trial is to determine if the long-term outcomes of patients who receive medical management for symptoms (e.g., headache, seizures) associated with an unruptured BAVM are superior to those who receive medical management and invasive therapy to eradicate the BAVM.

Participants will be randomly assigned to receive either symptomatic medical management alone or such management with invasive therapies (any combination of surgery, endovascular embolization, or radiotherapy). Functional assessment will be carried out at the time of randomization, pre-intervention and 48-hour post-intervention, and for all participants at 1 month, and at 6 month intervals throughout the follow up period which will be a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have unruptured BAVM diagnosed by MRI/MRA, CTA and/or angiogram
2. Patient must be 18 years of age or older
3. Patient must have signed Informed Consent, Release of Medical Information, and Health Insurance Portability and Accountability Act (HIPAA/U.S. only) Forms

Exclusion Criteria:

1. Patient has BAVM presenting with evidence of recent or prior hemorrhage
2. Patient has received prior BAVM therapy (endovascular, surgical, radiotherapy)
3. Patient has BAVM deemed untreatable by local team, or has concomitant vascular or brain disease that interferes with/or contraindicates any interventional therapy type (stenosis/occlusion of neck artery, prior brain surgery/radiation for other reasons)
4. Patient has baseline Rankin ≥2
5. Patient has concomitant disease reducing life expectancy to less than 10 years
6. Patient has thrombocytopenia (< 100,000/μL),
7. Patient has uncorrectable coagulopathy (INR>1.5)
8. Patient is pregnant or lactating
9. Patient has known allergy against iodine contrast agents
10. Patient has multiple-foci BAVMs
11. Patient has any form of arteriovenous or spinal fistulas

    Previous diagnosis of any of the following -
12. Patient has a diagnosed Vein of Galen type malformation
13. Patient has a diagnosed cavernous malformation
14. Patient has a diagnosed dural arteriovenous fistula
15. Patient has a diagnosed venous malformation
16. Patient has a diagnosed neurocutaneous syndrome such as cerebro-retinal angiomatosis (von Hippel-Lindau), encephalo-trigeminal syndrome (Sturge-Weber), or Wyburn-Mason syndrome
17. Patient has diagnosed BAVMs in context of moya-moya-type changes
18. Patient has diagnosed hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2006-10; Primary Completion 2013-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Difference of 5-year event rates between two arms | 5 years
  The hypothesis to be tested is that there is no difference between medical management and interventional therapy in the time to stroke or death from any cause.

SECONDARY OUTCOMES:
Prevalence of the risk of death or clinical impairment at 5 years post-randomization with early intervention | 5 years
  The hypothesis to be tested is that early intervention decreases the risk of death or clinical impairment at 5 years post-randomization. (Rankin Score >/= 2)

CONTACTS AND LOCATIONS:
Overall Officials: J.P. Mohr, MS, MD, Principal Investigator — Stroke Center/The Neurological Institute, Columbia University; Alan J. Moskowitz, MD, Principal Investigator — InCHOIR, Department of Health Policy, Mount Sinai School of Medicine; Michael Parides, PhD, Principal Investigator — InCHOIR, Department of Health Policy, Mount Sinai School of Medicine, Co-PI; Christian Stapf, MD, Principal Investigator — Clinical Coordinating Center, Europe; Eric Vicaut, MD, Principal Investigator — Clinical Coordinating Center, Europe, Co-PI; Claudia S. Moy, PhD, Principal Investigator — NINDS, Co-PI
Locations (66):
- United States (25):
  - Barrow Neurological Institute, 350 West Thomas Road, Phoenix, Arizona
  - Kaiser Permanente Los Angeles Medical Center,4867 Sunset Blvd, Los Angeles, California
  - University of California at Los Angeles, UCLA School of Medicine, 710 Westwood Plaza, Los Angeles, California
  - Kaiser Permanente (SF), Redwood City, California
  - University of California at San Francisco, 1001 Potrero Avenue- Rm 3C-38, San Francisco, California
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Stritch School of Medicine, Department of Neurology, 2160 S 1st Ave, Bldg 105/2700, Maywood, Illinois
  - University of Iowa Hospitals, Department of Neurology, 200 Hawkins Drive ,, Iowa City, Iowa
  - Michigan Head and Spine Institute, Providence Hospital and Medical Center, 16001 West Nine Mile Road, Southfield, Michigan
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - SUNY Downstate Medical Center, 451 Clarkson Avenue, Box 1189, Brooklyn, New York
  - Mercy Hospital of Buffalo, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, One Gustave L. Levy Place, Department of Neurosurgery- Box 1136, New York, New York
  - New York Presbyterian Hospital, Columbia Campus, Neurological Institute, 710 W. 168th St, New York, New York
  - John P. Murtha Neuroscience & Pain Institute,1450 Scapl Ave, Suite 120,, Johnstown, Pennsylvania
  - Thomas Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - Brackenridge Hospital, Brain and Spine Center, 601 East 15th Street, Austin, Texas
  - University of Texas Medical School in Houston, Houston, Texas
  - University of Virginia School of Medicine, Department of Neurosurgery, P.O. Box 800212, Charlottesville, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Wesley Medical Center, Auchenflower, Queensland
  - Austin Health, University of Melbourne 300 Waterdale Rd,Heidelberg Heights, Melbourne, Victoria
- Austria (2):
  - Universitätsklinik für Neurologie, Anichstrasse 35, 6020 Innsbruck, Innsbruck
  - Rudolfstiftung, Neurochirurgie, Juchgasse 25, A-1030, Vienna
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- Canada (3):
  - Hamilton General Hospital .237 Barton Street East, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - CHUM Notre Dame Hospital, Department of Radiology, 1560 Sherbrooke Street, Montreal, Quebec
- Helsinki University Central Hospital, Dept. of Neurosurgery, Topeliuksenkatu 5, Helsinki, P.O. Box 266, Helsinki, Finland
- France (6):
  - Hôpital de la Cavale-Blanche, Service de Neurologie, Bd. Tanguy Pringent, Brest
  - CHU Henri Mondor, Service de Neuroradiologie, Créteil
  - Centre Hospitalier Régional et Universitaire de Lille, Clinique de Neurochirurgie, Hopital Roger Salengro, CHRU, Lille
  - Hôpital Sainte Anne, Service de Neurochirurgie, Centre Hospitalier Sainte Anne, 1, Rue Cabanis, Paris
  - Hôpital Lariboisière, Service de Neuroradiologie, 2, Rue Ambroise Paré, Paris
  - European Coordinating Center: Dept. of Neurology, Hôpital Lariboisière, 2 Rue Ambroise Paré, 75475 Paris cedex 10,, Paris
- Germany (9):
  - Charité Campus Benjamin Franklin (CCBF), Neurologische Klinik, Hindenburgdamm 30, Berlin
  - Uniklinikum Dresden, Neuroradiologie, Fetscherstr. 74, Dresden
  - Universitätsklinikum Essen, Institut für Diagnostische und Interventionelle Radiologie und Neuroradiologie, Hufelandstraße 55, Essen
  - Uniklinikum Frankfurt, Institut für Neuroradiologie, Schleusenweg 2-16, Frankfurt am Main
  - Uniklinik Freiburg, Neuroradiology-Neurocenter, Breisacher Str. 64, Freiburg im Breisgau
  - Berufsgenossenschaftliche Kliniken Bergmannstrost, Klinik für Neurochirurgie, Merseburger Str. 165, Halle
  - Department of Neuroradiology, University Medical Center Hamburg-Eppendorf, Martinistrasse 52, Hamburg
  - Universitätsklinik Heidelberg, Department of Neurosurgery, Im Neuenheimer Feld 400, Heidelberg
  - Klinikum Großhadern, LMU München, Neurologische Klinik und Poliklinik, Marchionistr. 15, Munich
- Italy (2):
  - Bellaria Hospital, Department of Neurosurgery, Bologna
  - Servizio di Neuroradiologia, Ospedale San Raffaele, Via Olgettina 60, Milan
- Netherlands (2):
  - Department of Neurosurgery, Universitair Medisch Centrum Groningen Hanzeplein 1, Groningen
  - Utrecht University Hospital, Heidelberglaan 100, 3584 CX, Utrecht
- Seoul National University Hospital, Seoul, Seoul, South Korea
- Hospital Universitari de Bellvitge, Sección de Neuroradiologia, c/ Feixa Llarga s/n, L'Hospitalet de Llobregat, Barcelona, Spain
- Inselspital, Neurologische Klinik, 3010 Bern, Schweiz, Switzerland
- United Kingdom (10):
  - Frenchay Hospital, Neuroradiology Department, Bristol
  - Western General Hospital, Bramwell Dott Building, Department of Clinical Neurosciences, Crewe Road, Edinburgh
  - Consultant Neurologist, Department of Neurology, Leeds General Infirmary, Great George Street, Leeds
  - Walton Centre for Neurology, Lower Lane Fazakerley, Liverpool
  - Institute of Neurology, Box 6, The National Hospital, Queen Square, London
  - Department of Neurosurgery, Newcastle General Hospital, Westgate Road, Newcastle upon Tyne
  - Imaging Directorate, Derriford Hospital, Plymouth
  - Neuroscience Department, Royal Preston Hospital, Sharoe Green Lane, Fulwood, Preston
  - Department of Neurology, Hope Hospital, Salford
  - Department of Neurology, Royal Hallamshire Hospital, Glossop Road, Sheffield

REFERENCES:
- [Background] Stapf C, Mohr JP, Choi JH, Hartmann A, Mast H. Invasive treatment of unruptured brain arteriovenous malformations is experimental therapy. Curr Opin Neurol. 2006 Feb;19(1):63-8. doi: 10.1097/01.wco.0000200546.14668.78. PMID 16415679
- [Derived] Mohr JP, Overbey JR, Hartmann A, Kummer RV, Al-Shahi Salman R, Kim H, van der Worp HB, Parides MK, Stefani MA, Houdart E, Libman R, Pile-Spellman J, Harkness K, Cordonnier C, Moquete E, Biondi A, Klijn CJM, Stapf C, Moskowitz AJ; ARUBA co-investigators. Medical management with interventional therapy versus medical management alone for unruptured brain arteriovenous malformations (ARUBA): final follow-up of a multicentre, non-blinded, randomised controlled trial. Lancet Neurol. 2020 Jul;19(7):573-581. doi: 10.1016/S1474-4422(20)30181-2. PMID 32562682
- [Derived] Mohr JP, Overbey JR, von Kummer R, Stefani MA, Libman R, Stapf C, Parides MK, Pile-Spellman J, Moquete E, Moy CS, Vicaut E, Moskowitz AJ, Harkness K, Cordonnier C, Biondi A, Houdart E, Berkefeld J, Klijn CJM, Barreau X, Kim H, Hartmann A; International ARUBA Investigators. Functional impairments for outcomes in a randomized trial of unruptured brain AVMs. Neurology. 2017 Oct 3;89(14):1499-1506. doi: 10.1212/WNL.0000000000004532. Epub 2017 Sep 6. PMID 28878048
- [Derived] Mohr JP, Parides MK, Stapf C, Moquete E, Moy CS, Overbey JR, Al-Shahi Salman R, Vicaut E, Young WL, Houdart E, Cordonnier C, Stefani MA, Hartmann A, von Kummer R, Biondi A, Berkefeld J, Klijn CJ, Harkness K, Libman R, Barreau X, Moskowitz AJ; international ARUBA investigators. Medical management with or without interventional therapy for unruptured brain arteriovenous malformations (ARUBA): a multicentre, non-blinded, randomised trial. Lancet. 2014 Feb 15;383(9917):614-21. doi: 10.1016/S0140-6736(13)62302-8. Epub 2013 Nov 20. PMID 24268105
- [Derived] Stapf C. The rationale behind "A Randomized Trial of Unruptured Brain AVMs" (ARUBA). Acta Neurochir Suppl. 2010;107:83-5. doi: 10.1007/978-3-211-99373-6_13. PMID 19953376
- [Derived] Stapf C, Mohr JP. Unruptured brain arteriovenous malformations should be treated conservatively: yes. Stroke. 2007 Dec;38(12):3308-9. doi: 10.1161/STROKEAHA.107.504605. Epub 2007 Oct 25. No abstract available. PMID 17962585
- See also: An ARUBA web site has been developed to allow physicians to have access to up-to-date trial information. It will also be available to patients and their families. — http://www.arubastudy.org